CLINICAL TRIAL: NCT05948475
Title: A Phase III, Randomized, Controlled, Global Multicenter Study to Evaluate the Efficacy and Safety of Oral Tinengotinib VS Physician's Choice in Subjects With FGFR-altered, Chemotherapy- and FGFR Inhibitor-Cholangiocarcinoma
Brief Title: Study of Tinengotinib VS. Physician's Choice a Treatment of Subjects With FGFR-altered in Cholangiocarcinoma
Acronym: FIRST-308
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: TransThera Sciences (Nanjing), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TT420C2308
Record Dates: First submitted 2023-06-29; First posted 2023-07-17 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-05

CONDITIONS: Cholangiocarcinoma
Keywords: Refractory/Relapsed Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tinengotinib 8 mg QD (Experimental): Tinengotinib will be administered in 28-day cycles.
  Interventions: Drug: Tinengotinib 8 mg
- Tinengotinib 10 mg QD (Experimental): Tinengotinib will be administered in 28-day cycles.
  Interventions: Drug: Tinengotinib 10 mg
- Physician's Choice (Active Comparator): Physician's Choice treatments include FOLFOX or FOLFIRI
  Interventions: Drug: Physician's Choice

INTERVENTIONS:
Drug: Tinengotinib 8 mg — Subjects randomized to receive tinengotinib will receive a starting dose of either 8 mg QD., self-administered orally QD in 28-day cycles.
  Arms: Tinengotinib 8 mg QD
Drug: Tinengotinib 10 mg — Subjects randomized to receive tinengotinib will receive a starting dose of either10 mg QD., self-administered orally QD in 28-day cycles.
  Arms: Tinengotinib 10 mg QD
Drug: Physician's Choice — For subjects receiving FOLFOX or FOLFIRI, the subject will receive treatment every two weeks, with two administrations per each 28-day cycle.
  Arms: Physician's Choice

SUMMARY:
This study is a Phase III, Randomized, Controlled, Global Multicenter Study to Evaluate the Efficacy and Safety of Oral Tinengotinib versus Physician's Choice in Subjects with Fibroblast Growth Factor Receptor (FGFR)-altered, Chemotherapy- and FGFR Inhibitor-Refractory/Relapsed Cholangiocarcinoma

DETAILED DESCRIPTION:
Approximately 200 subjects will be enrolled. Eligible subjects will be randomized in a 2:2:1 ratio to receive tinengotinib 8 mg QD, tinengotinib 10 mg QD or Physician's Choice in Part A; and eligible subjects will be randomized in a 2:1 ratio to receive the recommended Part B dose or selected dose or Physician's Choice in Part B.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of signing the informed consent form (ICF).
2. Histologically or cytologically confirmed CCA/adenocarcinoma of biliary origin with radiological evidence of unresectable or metastatic disease.
3. Documentation of FGFR2 fusion/rearrangement gene status
4. Subjects must have received at least one line of prior chemotherapy and exactly one FDA approved FGFR inhibitor.

Exclusion Criteria:

1. Prior receipt of two or more FGFR inhibitors, either approved or investigational drugs.
2. Subjects with known brain or central nervous system (CNS) metastases that have radiologically or clinically progressed in the 28 days prior to initiation of therapy. Subjects with asymptomatic brain/CNS metastases or treated brain/CNS metastases that have been clinically stable for 14 days on steroids without escalation of steroids are eligible for enrollment.
3. Subjects with a known concurrent malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy, including those that have previously undergone potentially curative therapy.
4. Subjects who have received prior systemic therapy or investigational study drug ≤ 5 half-lives or 14 days, whichever is shorter, prior to starting the study drug or who have not recovered (grade ≤ 1 or at pretreatment baseline except tolerable grade 2 alopecia, fatigue/asthenia, and neuropathy due to trauma) from adverse events (AEs) of prior therapy.
5. Concurrent anticancer therapy including chemo-, immune-, or radiotherapy. Hormone therapy may be allowed with Sponsor approval.
6. Subjects who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting the study drug or who have not recovered from AEs of prior therapy.
7. Subjects with uncontrolled hypertension (defined as blood pressure of ≥ 150 mm Hg systolic and/or ≥ 90 mm Hg diastolic despite adequate treatment with antihypertensive medications at screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Part A: Incidence, duration, and severity of adverse events (AEs) | Up to 30 days from study discontinuation
  As assessed per Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (or the most current version).
Part B: PFS by BICR | From first study drug administration until the date of first documented progression assessed by BICR or date of death from any cause, whichever came first, assessed up to 24 months
  Progression-free survival (PFS) by BICR: PFS is defined as the time from date of randomization to the date of first documented disease progression as assessed by BICR per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or date of death due to any cause, whichever is earlier.

SECONDARY OUTCOMES:
Part A: ORR by Investigator | Through study completion, an average of 9 months.
  ORR:objective response rate (ORR), the proportion of subjects who achieved a complete response (CR) or a partial response (PR) based on RECIST version 1.1.
Part A: DOR by Investigator | Through study completion, an average of 9 months.
  Duration of response for CR or PR based on RECIST version 1.1.
Part B:Overall Survival (OS) | From first study drug administration until the date of death from any cause, assessed up to 24 months.
  OS is defined as the time from date of randomization to date of death of any cause.
Part B: Objective Response Rate (ORR) by BICR and by Investigator: | Through study completion, an average of 9 months.
  The proportion of subjects who achieved a complete response (CR) or a partial response (PR) based on RECIST version 1.1.
Part B: Duration of Response (DOR) by BICR and by Investigator | Through study completion, an average of 9 months.
  Duration of response for CR or PR based on RECIST version 1.1.
Part B: PFS by Investigators per RECIST v1.1. | From first study drug administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  PFS is defined as the time from date of randomization to the date of first documented disease progression as assessed by BICR per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Milind Javle, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (87):
- United States (19):
  - UCLA Medical Center, Santa Monica, California
  - Stanford Cancer Center, Stanford, California
  - The University of Kansas Cancer Center, Westwood, Los Angeles, California
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - The University of Chicago Hospitals, Chicago, Illinois
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford, Detroit, Michigan
  - University of Minnesota- Masonic Cancer Center, M Health Fairview, Minneapolis, Minnesota
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Messino Cancer Centers, Asheville, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Tennessee Oncology- Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Oncology-Sammons Cancer Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Austria (2):
  - Ordensklinikum Linz GmbH, Linz
  - Landesklinikum Wiener Neustadt, Wiener Neustadt
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
- France (8):
  - Institut Sainte Catherine - Institut du Cancer Avignon Provence, Avignon
  - Centre Hospitalier Régional Universitaire de Besançon, Besançon
  - Hopital Beaujon, Clichy
  - Hopital Franco-Britannique - Fondation Cognacq-Jay, Levallois-Perret
  - Clinique de la Sauvegarde, Lyon
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Hopital Saint Antoine, Paris
  - Institut de Cancerologie Gustave Roussy, Villejuif
- Germany (6):
  - Krebszentrum Reutlingen, Baden
  - Krankenhaus Nordwest gGmbH, Frankfurt
  - Asklepios Klinik Altona, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Heidelberg (UKHD) - Nationales Centrum fuer Tumorerkrankungen Heidelberg (NCT), Heidelberg
  - Ludwig-Maximilians-Universität München Kum, München
- Italy (13):
  - Clinica Oncologica, Ospedali Riuniti Umberto 1, Ancona
  - Candiolo Cancer Institute - FPO IRCCS, Candiolo
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Istituto Europeo di Oncologia IRCCS, Milan
  - ASST Grande Ospedale Metropolitano Niguard, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli, Napoli
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - Azienda Ospedaliera Universitaria di Parma, Parma
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Humanitas Research Hospital, Rozzano
  - Azienda Ospedaliera Universitaria Senese Policlinico Le Scotte, Siena
  - AOUI Verona - Ospedale Borgo Roma, Verona
- Amsterdam UMC, location AMC, Amsterdam, Netherlands
- Centrum Onkologii-Instytut im. Marii Skłodowskiej-Curie, Warsaw, Poland
- Portugal (2):
  - Centro Hospitalar Lisboa Norte CHLN EPE - Hospital de Santa Maria, Lisbon
  - Fundação Champalimaud, Lisbon
- South Korea (11):
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Inje University Haeundae Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (12):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitari Vall d´Hebron, Barcelona
  - Hospital Universitario Reina Sofa, Córdoba
  - Clinica Universidad de Navarra, Madrid
  - HM Hospital Universitario Madrid Sanchinarro - CIOCC, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de octubre, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital CGMH - Kaohsiung Branch, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (4):
  - Royal Marsden Hospital NHS, London
  - UCG-1st floor central, London
  - The Christie NHS Foundation Trust - Christie Hospital, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: No